CLINICAL TRIAL: NCT05372952
Title: An Investigator Initiated Trial to Evaluate the Safety and Feasibility of the DyNETIC-35 Cobalt Chromium Balloon-expandable Stent for the Treatment of Atherosclerotic Iliac Lesions Via a Trans-radial Approach - Bionetic-TRA
Brief Title: An Investigator Initiated Trial to Evaluate the Safety and Feasibility of the DyNETIC-35 Stent for Iliac Lesions Via a Trans-radial Approach
Status: Completed | Type: Observational
Sponsor: Klinikum Arnsberg (Other)
Responsible Party: Sponsor
Other Study IDs: ASL202201
Record Dates: First submitted 2022-05-02; First posted 2022-05-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Arterial Disease
Keywords: transradial access,
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dynetic-35 Peripheral Balloon-Expandable Stent System — Stenotic iliac lesions will be treated with the Dynetic 35 stent via a radial access

SUMMARY:
This feasibility study with a 30 day follow up period will assess the safety and feasibility of the Dynetic-35 stent for the treatment of peripheral iliac artery lesions via a trans-radial approach.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years
2. Subject is capable (no legally authorized representative allowed) to provide written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site prior to any study related procedure
3. Subject has provided written informed consent before any study specific test or procedure and is willing to comply with all protocol and follow-up requirements
4. Subjects have a target lesion(s) with ≥ 70% stenosis (visual estimate) located in the iliac arteries
5. Target lesion is a de novo, restenotic or occluded lesion
6. Reference lumen (vessel) diameter between 5mm and 10 mm
7. The target lesion can be successfully crossed with a guide wire
8. Patient is eligible for transradial access
9. Subject has symptomatic iliac artery disease defined as Rutherford category 2 or higher

Exclusion Criteria:

1. Subject is pregnant and/or breastfeeding or planning to become pregnant during the course of the study.
2. Subject is with a current medical condition with a life expectancy of less than one year.
3. Pre-existing target iliac artery aneurysm or perforation or dissection
4. Any medical condition that in the opinion of the investigator poses an unacceptable risk for implant of a stent according to the study indications like, sensitivity to metal ions, intolerance to contrast or antiplatelet, anticoagulant or thrombolytic medications required per the protocol
5. Abdominal aortic aneurysm (AAA) contiguous to the iliac artery target lesion requiring treatment
6. The subject is currently participating in an investigational drug, biologic, or another device study and has not reached their primary endpoint yet
7. Subjects with small diameter upper extremity arteries that posed a contraindication to the use of 6F sheath
8. Severe stenosis or calcification of upper extremity arteries
9. Patient height precluding transradial access with a 170 cm long catheter shaft
10. Patient with a history of aortic arch atheroembolism
11. Infrainguinal outflow lesions that need to be treated during the same index procedure
12. Patients with negative bilateral Allen or barbeau tests (Note: vascular access should be done via the left hand where possible)
13. Subject has IFU listed contraindication(s)
14. Subject has in-stent restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from vascular center of the clinic.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Access site complications | 1 hour post procedure
  bleeding, , pseudoaneurysm, arteriovenous fistula (AVF), radial artery rupture or occlusion
Stroke | 30 days
Death | 30 days
Transradial technical success | Immediately after stent placement via radial access
  Successful delivery of the Dynetic-35 stent at the lesion site with residual stenosis of ≤ 30%
Number of patients converting to femoral artery access | 1 hour post procedure
  Transradial access feasibility is assessed as number of patients in whom access is converted to femoral artery access due to failure to access the lesion via the radial artery

SECONDARY OUTCOMES:
Length of hospital stay [hours] | up to 30 days
Procedure time [min] | Intraoperative
Procedure cost | 1 hour post procedure
  Number and details of auxiliary devices and medication used
Time to ambulation | up to 30 days
  Time between patient left the cath lab/operating theatre, and patient was able to walk 100 meters and the access site remained stable
Patient satisfaction regarding access site | 24 hours post procedure
  Patient questionnaire assessing 8 questions (anxiety about the procedure, overall pain, back pain, difficulties in toiletting, walking, daily movement, selfcare and using the dominant hand) on a numeric rating scale (NRS, 0-10, 0 = none, 10 most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Lichtenberg, MD, Principal Investigator — Klinikum Hochsauerland GmbH
Locations (1):
- Vascular center of Klinikum Hochsauerland GmbH, Arnsberg, Germany